CLINICAL TRIAL: NCT06750926
Title: Optimal Position of the Third Generation Video Laryngeal Mask Airway: to Compare Visualization of the SaCoVLMTM Videoscope With the Traditional Fiberoptic Bronchoscope
Brief Title: Optimizing Third-Generation Video Laryngeal Mask Position: SaCoVLM™ vs. Fiberoptic Bronchoscope
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KMUHIRB-F(II)-20240241
Record Dates: First submitted 2024-12-18; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Supraglottic Airway Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients placed SaCoVLM checked position by real-time video image (Experimental): patients placed SaCoVLM checked position by real-time video image, including native camera and fiberoptic endoscopy
  Interventions: Diagnostic Test: video image through laryngeal mask specific channel

INTERVENTIONS:
Diagnostic Test: video image through laryngeal mask specific channel — patients placed SaCoVLM will be checked the proper position of placement by native camera through specific video channel and fiberoptic endoscopy through ventilation channel perspectively

SUMMARY:
This study aims to compare the effectiveness of SaCoVLM™ in artificial airway ventilation during general anesthesia, focusing on the correlation between native video camera imaging and fiberoptic endoscopy. Primary outcomes include the analysis of imaging correlation, while secondary outcomes assess initial placement success rates, difficulty, blood clot adherence, vital sign changes, and postoperative complications.

DETAILED DESCRIPTION:
In modern medicine, the management of artificial airways is a crucial component of patient care in emergency departments, operating rooms, and intensive care units, where it plays a vital role in providing respiratory ventilation. The laryngeal mask airway (LMA) is a type of supraglottic airway device. Due to its ease of placement and improvements in ventilation seal and overall angle design, it is now widely used in various clinical situations and can even replace some functions of endotracheal intubation.

However, despite the LMA's ease of placement, operators with limited experience often struggle to adjust it to the optimal position, significantly impacting ventilation effectiveness. Traditionally, to confirm the correct placement of the LMA, practitioners rely on both experiential physical examinations and objective data such as capnography waveforms, leak pressure measurements, ultrasound, and fiberoptic endoscopy images.

The SaCoVLM™ video laryngeal mask is a third-generation supraglottic device that integrates an imaging system, allowing for real-time lateral video recording during placement to observe the relative position of the LMA tip with respect to the vocal cords and surrounding structures.

The aim of this study is to compare the use of SaCoVLM™ for artificial airway ventilation during routine surgical general anesthesia, specifically evaluating the placement adjustments using two different imaging perspectives: the native video camera and fiberoptic endoscopy. The primary outcome is the analysis of the correlation between the two types of imaging. Secondary outcomes include the success rate and difficulty of initial placement of the SaCoVLM™, whether visible blood clots adhere to the device upon removal, changes in vital signs before and after placement, and postoperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I~III, age 18~65 y/o, BMI 18~30kg/m2, elective surgery, surgery duration < 2 hours, supine position, general anesthesia with laryngeal mask airway insertion

Exclusion Criteria:

* Smoking, betel nuts use, any known anatomical variation or disease of facial or airway structure, anticipated difficult airway, limited mouth opening distance or neck motility, loosening teeth, gastroesophageal reflux history, ongoing upper airway infection or inflammation symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
correlation of native camera image of SaCoVLM and traditional fiberoptic endoscopy image | From enrollment to postoperative day 1
  The primary outcome is the analysis of the correlation between the two types of imaging, native camera image of SaCoVLM and traditional fiberoptic endoscopy image, to confirm proper position of laryngeal mask placement.

SECONDARY OUTCOMES:
the success rate and difficulty of initial placement of the SaCoVLM™ | From enrollment to postoperative day 1
  One of the secondary outcomes is the success rate and difficulty of initial placement of the SaCoVLM™. We will record the number of attempts to place or adjust the laryngeal mask to proper position.
whether visible blood clots adhere to the device upon removal | From enrollment to postoperative day 1
  One of the secondary outcomes is whether visible blood clots adhere to the device upon removal.
changes in heart rate values before and after SaCoVLM placement | From enrollment to postoperative day 1
  One of the secondary outcomes is changes in heart rate values before and after SaCoVLM placement.
changes in mean arterial blood pressure values before and after SaCoVLM placement | From enrollment to postoperative day 1
  One of the secondary outcomes is changes in mean arterial blood pressure values before and after SaCoVLM placement.
postoperative adverse events | From enrollment to postoperative day 1
  One of the secondary outcomes is postoperative adverse events such as sore throat, pain on swallowing, hoarseness, numbness of the tongue, or jaw pain. We will record all the events above along with their severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided